CLINICAL TRIAL: NCT06868446
Title: Dosage, Feasibility, Acceptability and Usability of OTX-601
Brief Title: Feasibility of a Digital Therapeutic for Adults With Posttraumatic Stress Disorder (PTSD)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oui Therapeutics, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 2024-Oui-002; R44MH136888 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: PTSD; Post Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OTX-601 Version 1 (Experimental): A prescription digital therapeutic designed to overcome existing barriers and deliver evidence-based treatment for PTSD
  Interventions: Device: Digital Therapeutic (Version 1); Behavioral: Treatment as Usual (TAU)
- OTX-601 Version 2 (Experimental): Increased dose of a prescription digital therapeutic designed to overcome existing barriers and deliver evidence-based treatment for PTSD
  Interventions: Device: Digital Therapeutic (Version 2); Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Device: Digital Therapeutic (Version 1) — Prescription digital therapeutic designed to overcome existing barriers and deliver evidence-based treatment for PTSD
  Arms: OTX-601 Version 1
Device: Digital Therapeutic (Version 2) — Prescription digital therapeutic (increased dose) designed to overcome existing barriers and deliver evidence-based treatment for PTSD
  Arms: OTX-601 Version 2
Behavioral: Treatment as Usual (TAU) — Treatment as usual may include psychotherapy and/or pharmacological interventions.

SUMMARY:
This study is exploring the efficacy of a digital therapeutic app in reducing symptoms of posttraumatic stress disorder (PTSD) in adults.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a randomized controlled trial to evaluate the usability and feasibility as well as the safety and effectiveness of OTX-601 (version 1) + TAU compared to OTX-601 (version 2) + TAU in reducing PTSD symptoms from baseline to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Posttraumatic stress disorder (PTSD) diagnosis
* Anxiety Sensitivity Index 3 (ASI-3) scores above 24
* PTSD Checklist for DSM-V (PCL-5) scores above 30
* Understands and speaks English
* Access to a smartphone that is connected to the internet

Exclusion Criteria:

* Score of 24 or lower on the ASI-3
* Score of 30 and below on the PCL-5
* No PTSD diagnosis
* Active psychosis
* Acute intoxication during study baseline
* Enrolled in another treatment research study
* Medical illness that would prevent the completion of interoceptive exposure exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-V (PCL-5) | Baseline, week 1, week 2, week 3, and week 7
  Change in PTSD symptoms will be ascertained with the PTSD Checklist for DSM-V (PCL-5). The PCL-5 total score ranges from 0 to 80, with higher scores indicating more severe symptoms.
System Usability Scale (SUS) | week 1, week 2, and week 3
  App usability will be ascertained with the System Usability Scale (SUS). The SUS provides a score from 0 to 100. An average SUS score equal to or greater than 68 is considered usable.

SECONDARY OUTCOMES:
Anxiety Sensitivity Index 3 (ASI-3) | Baseline, week 1, week 2, week 3 and week 7
  Change in anxiety sensitivity level will be ascertained with the Anxiety Sensitivity Index 3 (ASI-3). The ASI-3 total score ranges from 0 to 72 with a higher score indicating greater anxiety sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Simon, PhD, Principal Investigator — Oui Therapeutics, Inc.